CLINICAL TRIAL: NCT03046875
Title: The Biophysical Impact of Transcutaneous Spinal Cord Stimulation Within a Single Session
Acronym: TSCS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never initiated because of lack of funding and research priorities have been shifted elsewhere.
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, Rebecca Martin, OTR/L, OTD, Manager Clinical Education and Training, International Center for Spinal Cord Injury Assistant Professor, Johns Hopkins School of Medicine, Dept. of Physical Medicine and Rehabilitation, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00103592
Record Dates: First submitted 2017-02-02; First posted 2017-02-08 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcutaneous Spinal Cord Stimulation (Experimental): Subjects will participate in a single session of Transcutaneous Spinal Cord Stimulation, involving 30 minutes of stimulation with isokinetic strength testing of knee extension.
  Interventions: Other: Transcutaneous Spinal Cord Stimulation
- Sham (Sham Comparator): Subjects will participate in a single session of isokinetic strength testing of knee extension with sham stimulation.
  Interventions: Other: Sham stimulation

INTERVENTIONS:
Other: Transcutaneous Spinal Cord Stimulation — Transcutaneous Spinal Cord Stimulation is a non-invasive mechanism to enhance excitation of spinal neural circuitry and represents a promising supplement to existing physical therapy programs. Transcutaneous Spinal Cord Stimulation will be applied (via the Vectra Neo) using a 5cm x10cm oval electrode placed midline on the skin between spinous process T11 -T12 as a cathode and two 7.5cm x 13cm rectangular electrodes placed symmetrically on the skin over the lower abdomen as anodes.7,9 A symmetrical biphasic rectangular waveform, at 50Hz and 1millisecond, will be used to provide 30 continuous minutes of stimulation.
  Other Names: TSCS
  Arms: Transcutaneous Spinal Cord Stimulation
Other: Sham stimulation — Sham procedures, well documented in Transcranial DC Stimulation (tDCS), will be used. Electrodes will be placed as they are in the Transcutaneous Spinal Cord Stimulation condition. Stimulation will be applied at subject's maximum intensity for 30 seconds and then discontinued.
  Arms: Sham

SUMMARY:
To determine the biophysical impact of biophysical Impact of Transcutaneous Spinal Cord Stimulation (TSCS) within a single session. We hypothesize that subjects will demonstrate increased volitional muscle strength with TSCS. This will be assessed by isokinetic strength testing of post-injury dominant-side knee extension. Subjects will be tested in both Transcutaneous Spinal Cord Stimulation and sham conditions.

DETAILED DESCRIPTION:
The investigators will conduct isokinetic strength testing (via the Biodex) of post-injury, dominant-side knee extension before, during, and after TSCS and a sham condition. Transcutaneous Spinal Cord Stimulation will be applied (via the Vectra Neo) using a 5cm x10cm oval electrode placed midline on the skin between spinous process T11 -T12 as a cathode and two 7.5cm x 13cm rectangular electrodes placed symmetrically on the skin over the lower abdomen as anodes. A symmetrical biphasic rectangular waveform, at 50Hz and 1millisecond, will be used to provide 30 continuous minutes of stimulation. As sham procedures for this intervention have not been established, the investigators will follow sham procedures well documented in Transcranial DC Stimulation (tDCS). Electrodes will be placed as they are in the Transcutaneous Spinal Cord Stimulation condition. Stimulation will be applied at subject's maximum intensity for 30 seconds and then discontinued. Subjects will participate in two testing sessions, each approximately one hour in length, separated by at least 24 hours.

Subject's starting condition will be randomized. Subjects will be informed that two stimulation conditions are being tested, but will not be told which is the experimental condition.

ELIGIBILITY:
Inclusion Criteria:

* > 1 year post spinal cord injury
* Non-progressive spinal cord injury
* Neurological level above T10
* Tolerates upright position for >30 minutes
* Medically stable (no hospitalizations in last 3 months)
* Unilateral knee extension strength >/= 1/5 MMT
* Able to comply with procedures and follow up
* Are legally able to make their own health care decisions

Exclusion Criteria:

* Progressive SCI/D (MS, ALS, ADEM, etc.)
* Opens wounds at stimulation site
* Pregnant women
* ROM limits of >10 degree of knee flexion or extension
* Cardiac pacemaker/defibrillator
* Active cancer diagnosis
* Currently receiving TSCS
* Evidence of uncontrolled autonomic dysreflexia
* Non- English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Knee extension strength | Day 1, Day 2
  Change in isokinetic strength assessment of the post-injury dominant side quadripceps

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Martin, OTR/L, OTD, CPAM, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Rebecca Martin, OTR/L, OTD, CPAM, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No